CLINICAL TRIAL: NCT01098409
Title: Mechanisms of Nitrite Mediated Cardioprotection in Coronary Artery Bypass Surgery
Brief Title: Nitrite Mediated Cardioprotection During Coronary Artery Bypass Surgery
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Birmingham NHS Foundation Trust (Other)
Responsible Party: Professor Robert Bonser, University Hospitals Birmingham NHS Trust
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RRK3719; RG/04/005/14168 (Other Grant/Funding Number: British Heart Foundation); 09/H1207/7 (Other: South Birmingham Research and Ethics Committee)
Record Dates: First submitted 2010-03-30; First posted 2010-04-02 (Estimated); Last update posted 2010-04-02 (Estimated); Status verified 2010-01

CONDITIONS: Coronary Artery Bypass Surgery
Keywords: sodium nitrite; coronary artery bypass surgery; cardioprotection; myocardial injury
MeSH Terms: interventions — Sodium Nitrite; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- sodium nitrite 24 hours before (Experimental)
  Interventions: Drug: sodium nitrite
- sodium nitrite during surgery (Experimental)
  Interventions: Drug: sodium nitrite
- 0.9% sodium chloride (Placebo Comparator)
  Interventions: Drug: 0.9% sodium chloride

INTERVENTIONS:
Drug: sodium nitrite — 0.2mcg/kg/min or 1mcg/kg/min intravenous for 30minutes at 1ml/min
  Arms: sodium nitrite 24 hours before; sodium nitrite during surgery
Drug: 0.9% sodium chloride — intravenous 0.9% sodium chloride over 30minutes at 1ml/min
  Arms: 0.9% sodium chloride

SUMMARY:
The purpose of this study is to determine whether sodium nitrite administration 24 hours prior to or during coronary artery bypass surgery protects the heart better from lack of blood flow which occurs as part of this type of operation. The study will also determine what the mechanisms of this cardioprotection are.

DETAILED DESCRIPTION:
In recent years, there has been much interest in sodium nitrite as a cytoprotective agent in in vitro and animal models. A recent study undertaken in a canine model of myocardial infarction demonstrated a 50% reduction in myocardial injury following the administration of sodium nitrite prior to the ischemic event. In humans, the setting of coronary artery bypass surgery lends itself well to study potential cytoprotective agents. During cardiac surgery, the heart undergoes a period of ischemia allowing the surgeons to operate on the heart. This is followed by a period of reperfusion which in itself can add to cellular injury. Such injury can hinder post-operative myocardial recovery.

The aim of this pilot study is to determine whether the cardioprotective effects of sodium nitrite demonstrated in animal models are translated in humans and to determine the exact underlying mechanisms of this cytoprotection. Patients undergoing coronary artery bypass grafting surgery who give written, informed consent will receive sodium nitrite 24 hours prior to surgery, during cardiac surgery or placebo. Myocardial injury will be assessed through the measurement of biochemical markers such as troponin T. Cardiac biopsy samples will be obtained to determine underlying molecular mechanisms of this cardioprotection. The other aim of this pilot study is to determine what dose of sodium nitrite (i.e. 0.2mcg/kg/min or 1mcg/kg/min) is optimal for cardioprotection. This study will form pilot data also for a larger clinical trial with clinical endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective first time multi-vessel coronary artery bypass surgery
* Older than 18 years of age

Exclusion Criteria:

* Significant psychiatric /neurological impairment that might prevent adherence to the requirements of the protocol or the ability to give informed consent
* Inability to read the Information Sheet.
* Redo operation
* Age >80 years
* Pregnancy
* Renal Impairment requiring pre-operative renal support
* Diabetes Mellitus
* Intended heart valve or additional surgery
* Episodes of angina or ischemia within 48hours prior to the procedure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-02; Primary Completion 2012-01 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Troponin T | 72 hours post release of aortic cross clamp
  Biochemical marker of myocardial injury

SECONDARY OUTCOMES:
Troponin T | 6 hours post release of aortic cross clamp
troponin T | 12 hours post release of aortic cross clamp
Troponin T | 24 hours post release of aortic cross clamp
Troponin T | 48 hours post release of aortic cross clamp
Creatinine Kinase myocardial Fraction (CKMB) | 6 hours post release of aortic cross clamp
Creatinine Kinase myocardial Fraction (CKMB) | 12 hours post release of aortic cross clamp
Creatinine Kinase myocardial Fraction (CKMB) | 24 hours post release of aortic cross clamp
Creatinine Kinase myocardial Fraction (CKMB) | 48 hours post release of aortic cross clamp
Creatinine Kinase myocardial Fraction (CKMB) | 72 hours post release of aortic cross clamp
venous methemoglobinaemia | immediately before infusion of study drug
  study drug means both sodium nitrite and placebo
plasma 8-isoprostane | before aortic cross clamp administration
Nitric oxide metabolites in cardiac tissue | before aortic cross clamp application
Cardiac output studies | upto 12 hours after release of aortic cross clamp
inotrope usage | up to 12 hours after release of aortic cross clamp
venous methemoglobinemia | immediately after infusion of study drug.
  Study drug could be sodium nitrite or placebo and each infusion last 30minutes.
Nitric oxide metabolites in cardiac tissue | before release of aortic cross clamp
Nitric oxide metabolites in cardiac tissue | 10minutes after release of aortic cross clamp
Plasma 8 isoprostane levels | 5minutes after discontinuation of cardiopulmonary bypass

CONTACTS AND LOCATIONS:
Overall Officials: Michael P Frenneaux, MD, Principal Investigator — University of Aberdeen
Locations (1):
- University Hospitals Birmingham NHS Trust, Birmingham, United Kingdom